CLINICAL TRIAL: NCT05715476
Title: The Effect of Different Altitude Levels on Spinal Anesthesia in Cesarean Section Surgery; Comparison of Anesthesia Parameters and Hemodynamic Changes
Brief Title: The Effect of Different Altitude Levels on Spinal Anesthesia in Cesarean Section Surgery
Acronym: altitude
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, Dilek Yeniay, Anesthesiology and Reanimation physician, Giresun University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DYeniay
Record Dates: First submitted 2022-11-28; First posted 2023-02-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Pregnant; High Altitude
Keywords: high altitude; moderately altitude; cesarian; pregnant
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- sea levelaltitude (Active Comparator): Pregnant women living in Giresun(sea levelaltitude),Turkey and undergoing cesarean section under elective conditions.
  Interventions: Procedure: cesarian surgery
- moderate altitude (Active Comparator): Pregnant women living in Çorum(moderate altitude),Turkey and undergoing cesarean section under elective conditions.
  Interventions: Procedure: cesarian surgery
- high altitude (Active Comparator): Pregnant women living in Van(high altitude),Turkey and undergoing cesarean section under elective conditions.
  Interventions: Procedure: cesarian surgery

INTERVENTIONS:
Procedure: cesarian surgery — The same anesthesia protocol will be applied to the patient group at each altitude. In the sitting position, the spinal space was entered with a 25 gauge Quincke-tipped needle from the L4-5 space and a drop of CSF will be dripped onto the pH paper. Immediately afterwards, 12 mg of 0.5% hyperbaric bupivacaine will be given. The color formed on the pH paper will be noted. Sensory block level will be tested with pinprick test and motor block level will be evaluated with Modified Bromage scale. The number and duration of spinal anesthesia applications, the time of occurrence of sensory block in the T6 dermatome, the time to reach each score of the MB scale, the duration of the operation, the highest level of sensory block and anesthetic complications will be recorded. Sensory block time and motor block time of the patients followed in the service will be recorded.
  Other Names: sea level altitude, moderate altitude, high altitude

SUMMARY:
The aim of the researchers in this prospective study is to determine the differences, if any, in terms of anesthetic parameters among pregnant women who live at different altitudes and undergo cesarean section under neuraxial anesthesia under elective conditions and to contribute to the literature.

DETAILED DESCRIPTION:
Increased intra-abdominal pressure during pregnancy increases the pressure in the epidural and spinal space and causes enlargement of the epidural veins. This may lead to easier increases in the anesthetic blockage level. For this reason, it is necessary to use the lowest possible dose of local anesthesia in these individuals compared to normal healthy individuals.

The literature on the effect of altitude difference on central neuraxial block is limited. Based on studies showing changes in CSF volume and content in hypoxic conditions, According to the researchers, with the same amount of local anesthetic, the duration of sensory and motor blockade at sea level is thought to be equal to or longer than in mid-high regions.

This study will be carried out among pregnant women who live in the city center at 3 different altitudes [0-10 m (Giresun), 810 m (Çorum), 1725 m (Van)] and undergo cesarean section under elective conditions. It will be performed in a multicenter, prospective, controlled, randomized manner in order to determine the differences, if any, among these pregnant women in terms of anesthetic parameters.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years old
* Pregnant women 160-170 centimeters tall
* Be residing in the place of participation for at least 1 month

Exclusion Criteria:

* >ASA 2 pregnant women
* Contraindicated for spinal anesthesia, such as infection or coagulation disorder at the needle insertion site
* Pregnant women to be taken under emergency conditions

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant woman aged 18-40
Enrollment: 150 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
age | preoperative period
  18-40 age frame
Body max index | preoperative period
  kg/m2
heart rate | during the surgery
  beats/min
American Society of Anesthesiologists (ASA) | preoperative period
  ASA I and II
mean arterial pressure | during the surgery
  mmHg
The number and duration of spinal anesthesia applications | during the surgery
  second
the duration of sensory block formation in the T6 dermatome | during the surgery
  second
the time to reach each score of the MB(Modified bromage scale) scale 1-2-3 | during the surgery
  second
the duration of the operation (time from the beginning of the surgical incision to the completion of the surgery) | during the surgery
  minute
the highest level of sensory block | during the surgery
  dermatome level

SECONDARY OUTCOMES:
postoperative block parameters | postoperative first 24 hour
  Sensory block time (DBS) (time from local anesthetic injection until S2 dermatome sensation), motor block time (MBS) (time from local anesthetic injection to full motor function recovery) will be evaluated for the patients followed in the service.
postoperative headache parameter | postoperative first and 7. day
  On the first and seventh days after the operation, the patients will be questioned by the researcher for post-dural puncture headache (PDPH, increased pain intensity when standing up from the supine position) by phone call.
postoperative nausea and vomiting parameter | postoperative first 24 hour
  the degree of postoperative nausea and vomiting will be checked (Verbal Descriptive Scale).

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Yeniay, Principal Investigator — Giresun Universıty TURKEY
Locations (1):
- Gıresun gynecology and children's hospital, Giresun, Turkey (Türkiye)

REFERENCES:
- [Result] Leissner KB, Mahmood FU. Physiology and pathophysiology at high altitude: considerations for the anesthesiologist. J Anesth. 2009;23(4):543-53. doi: 10.1007/s00540-009-0787-7. Epub 2009 Nov 18. PMID 19921365
- [Result] Penaloza D, Arias-Stella J. The heart and pulmonary circulation at high altitudes: healthy highlanders and chronic mountain sickness. Circulation. 2007 Mar 6;115(9):1132-46. doi: 10.1161/CIRCULATIONAHA.106.624544. PMID 17339571
- [Result] Wilson MH, Edsell ME, Davagnanam I, Hirani SP, Martin DS, Levett DZ, Thornton JS, Golay X, Strycharczuk L, Newman SP, Montgomery HE, Grocott MP, Imray CH; Caudwell Xtreme Everest Research Group. Cerebral artery dilatation maintains cerebral oxygenation at extreme altitude and in acute hypoxia--an ultrasound and MRI study. J Cereb Blood Flow Metab. 2011 Oct;31(10):2019-29. doi: 10.1038/jcbfm.2011.81. Epub 2011 Jun 8. PMID 21654697
- [Result] Blayo MC, Coudert J, Pocidalo JJ. Ccomparison of cisternal and lumbar cerebrospinal fluid pH in high altitude natives. Pflugers Arch. 1975 Apr 29;356(2):159-67. doi: 10.1007/BF00584295. PMID 239384
- [Result] Sorensen SC, Milledge JS. Cerebrospinal fluid acid-base composition at high altitude. J Appl Physiol. 1971 Jul;31(1):28-30. doi: 10.1152/jappl.1971.31.1.28. No abstract available. PMID 5556959
- [Result] Carpenter RL, Hogan QH, Liu SS, Crane B, Moore J. Lumbosacral cerebrospinal fluid volume is the primary determinant of sensory block extent and duration during spinal anesthesia. Anesthesiology. 1998 Jul;89(1):24-9. doi: 10.1097/00000542-199807000-00007. PMID 9667290
- [Result] Hocking G, Wildsmith JA. Intrathecal drug spread. Br J Anaesth. 2004 Oct;93(4):568-78. doi: 10.1093/bja/aeh204. Epub 2004 Jun 25. No abstract available. PMID 15220175
- [Result] Aksoy M, Ince I, Ahiskalioglu A, Karaca O, Bayar F, Erdem AF. Spinal anaesthesia at low and moderately high altitudes: a comparison of anaesthetic parameters and hemodynamic changes. BMC Anesthesiol. 2015 Sep 10;15:123. doi: 10.1186/s12871-015-0104-y. PMID 26357836

DOCUMENTS (3):
  • Study Protocol (2023-01-25): https://cdn.clinicaltrials.gov/large-docs/76/NCT05715476/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT05715476/SAP_001.pdf
  • Informed Consent Form (2023-01-25): https://cdn.clinicaltrials.gov/large-docs/76/NCT05715476/ICF_002.pdf